CLINICAL TRIAL: NCT04048070
Title: Benefits of Enhanced Recovery After Surgery in Patients Undergoing Endoscopic Sinus Surgery
Brief Title: The Effect of Enhanced Recovery After Surgery in Endoscopic Sinus Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Principal Investigator, Luo Zhang, vise president of BeijingTongren Hospital, Beijing Tongren Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: TR-ERAS
Record Dates: First submitted 2019-08-05; First posted 2019-08-07 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Chronic Rhinosinusitis (Diagnosis); Surgery
MeSH Terms: conditions — Disease | interventions — flurbiprofen axetil; Sufentanil

STUDY DESIGN:
Intervention Model Description: Patients with chronic rhinosinusitis undergoing ESS were prospectively assigned to one of five groups; ERAS groups with postoperative intravenous Flubiprofen Axetil or analgesia pump, traditional care with Flubiprofen Axetil or analgesia pump (NERAS groups), or traditional care without postoperative intravenous analgesia group (control).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- ERAS with postoperative intravenous Flubiprofen Axetil (Experimental): The patients was given extended perioperative counseling, shorter fasting food for 6 to 8 hours and carbohydrate water for 2 hours before surgery. Early ambulation and oral intake 2 hours after patient recovery from anesthesia. Once a day 100mg Flubiprofen Axetil in this group for postoperative pain management.
  Interventions: Drug: Flurbiprofen Axetil; Behavioral: Extended perioperative counseling; Behavioral: Shorter fasting food and water time before surgery
- ERAS with analgesia pump (Experimental): The patients was given extended perioperative counseling, shorter fasting food for 6 to 8 hours and carbohydrate water for 2 hours before surgery. Early ambulation and oral intake 2 hours after patient recovery from anesthesia. An electronic analgesic pump containing opioids drug and Flubiprofen Axetil in this group for postoperative pain management.
  Interventions: Drug: Sufentanil; Behavioral: Extended perioperative counseling; Behavioral: Shorter fasting food and water time before surgery
- Traditional care with Flubiprofen Axetil (Experimental): Conventional perioperative counseling and regular fasting food for 12 hours and water for 6 hours before surgery. Lie down and oral intake at least 4 hours after recovery. Once a day 100mg Flubiprofen Axetil in this group for postoperative pain management.
  Interventions: Drug: Flurbiprofen Axetil; Behavioral: Conventional perioperative counseling; Behavioral: Regular fasting food and water time before surgery
- Traditional care with analgesia pump (Experimental): Conventional perioperative counseling and regular fasting food for 12 hours and water for 6 hours before surgery. Lie down and oral intake at least 4 hours after recovery. An electronic analgesic pump containing opioids drug and Flubiprofen Axetil in this group for postoperative pain management.
  Interventions: Drug: Sufentanil; Behavioral: Conventional perioperative counseling; Behavioral: Regular fasting food and water time before surgery
- traditional care without postoperative intravenous analgesia. (Placebo Comparator): Conventional perioperative counseling and regular fasting food for 12 hours and water for 6 hours before surgery. Lie down and oral intake at least 4 hours after recovery. Intravenous saline with necessary oral analgesic for postoperative pain management.
  Interventions: Behavioral: Conventional perioperative counseling; Behavioral: Regular fasting food and water time before surgery

INTERVENTIONS:
Drug: Flurbiprofen Axetil — One kind of NSAIDs, 200mg for 48 hours after surgery.
  Arms: ERAS with postoperative intravenous Flubiprofen Axetil; Traditional care with Flubiprofen Axetil
Drug: Sufentanil — One kind of opioid drugs, 1.5μg/kg, and recorded the drug consumption after surgery
  Arms: ERAS with analgesia pump; Traditional care with analgesia pump
Behavioral: Extended perioperative counseling — The extended perioperative counseling contained additional information, including surgery procedures, importance of medicine treatment and medical help to relieve depression and anxiety about disease during peri-operation period.
  Arms: ERAS with analgesia pump; ERAS with postoperative intravenous Flubiprofen Axetil
Behavioral: Shorter fasting food and water time before surgery — The patients in ERAS group were required to fast food for 6 to 8 hours and provided 12.6% maltodextrin carbohydrate supplement beverage for 2 hours before surgery
  Arms: ERAS with analgesia pump; ERAS with postoperative intravenous Flubiprofen Axetil
Behavioral: Conventional perioperative counseling — THe conventional perioperative counseling included the risk of surgery and prognosis of disease and other things patients need to know.
  Arms: Traditional care with Flubiprofen Axetil; Traditional care with analgesia pump; traditional care without postoperative intravenous analgesia.
Behavioral: Regular fasting food and water time before surgery — The stricter control of preoperative fasting requirements, prohibiting solids and liquids from previous midnight to operation time.
  Arms: Traditional care with Flubiprofen Axetil; Traditional care with analgesia pump; traditional care without postoperative intravenous analgesia.

SUMMARY:
Enhanced recovery after surgery (ERAS) protocols have been widely applied during perioperative periods for different diseases, there are few reports of ERAS in patients undergoing endoscopic sinus surgery (ESS). This study therefore aimed to evaluate the benefits of ERAS protocol compared to traditional care following ESS.

ELIGIBILITY:
Inclusion Criteria:

* The patient has CRSwNP need endoscopic sinus surgery for treatment.

Exclusion Criteria:

* age under 18 years
* pregnant
* ASA grade IV
* received oral or topical steroids within 4 weeks preceding surgery
* had previous ESS history
* intolerant to NSAIDS
* comorbidity of severe mental disease
* not compliant with therapy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2018-05-03 (Actual); Primary Completion 2018-10-15 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
Pain management | at 2 hours after surgery
  The pain scores after surgery were scored on a visual analogue scale of 0 to 10 as previously described, with 0 being no complaints whatsoever and 10 being the worst imaginable.
Pain management | at 6 hours after surgery
  The pain scores after surgery were scored on a visual analogue scale of 0 to 10 as previously described, with 0 being no complaints whatsoever and 10 being the worst imaginable.
Pain management | at 24 hours after surgery
  The pain scores after surgery were scored on a visual analogue scale of 0 to 10 as previously described, with 0 being no complaints whatsoever and 10 being the worst imaginable.
Pain management | at 48 hours after surgery
  The pain scores after surgery were scored on a visual analogue scale of 0 to 10 as previously described, with 0 being no complaints whatsoever and 10 being the worst imaginable.

SECONDARY OUTCOMES:
Hunger scores | at 5 minutes before surgery start
  The hunger scores before surgery were scored on a visual analogue scale of 0 to 10 as previously described, with 0 being no complaints whatsoever and 10 being the worst imaginable.
Self-rating Anxiety Scale | at baseline and 72 hours after surgery
  The anxiety scale was measured by Self-rating Anxiety Scale (SAS) questionaire. The SAS questionaire contain 20 items and each item is range 1 to 4 points. The total scores is reported, which range 20 to 80 points and higher scores mean that more anxiety.
thirst scores | at 5 minutes before surgery start
  The thirst scores before surgery were scored on a visual analogue scale of 0 to 10 as previously described, with 0 being no complaints whatsoever and 10 being the worst imaginable.
General comfort scores | at baseline and 72 hours after surgery
  Kolcaba General Comfort Questionnaire (GCQ) was assessed to evaluate the quality of life of patients. The GCQ questionaire contain 28 items and each item is range 1 to 4 points. The total scores is reported, which range 28 to 112 points and higher scores mean that feel more comfort.
quality of sleeping | at baseline and 72 hours after surgery
  Medical Outcomes Study Sleep Scale (MOS-SS) was assessed to evaluate the quality of sleep of patients. The MOS-SS questionaire contain 7 items, including sleep disturbance, snoring, awakening short of breath or with headache, sleep adequacy, daytime somnolence and amount of sleeping.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tongren Hospital, Beijing, Beijing Municipality, China